CLINICAL TRIAL: NCT01255787
Title: A Multinational, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Assess the Efficacy and Safety of Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: Efficacy and Safety Study of Vortioxetine (Lu AA21004) for Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004/CCT-002; 2010-022257-41 (EudraCT Number); U1111-1117-6595 (Registry Identifier: WHO); JapicCTI-101344 (Registry Identifier: JapicCTI); CTRI/2011/08/001963 (Registry Identifier: CTRI)
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Depression; Melancholia; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): Vortioxetine placebo-matching tablets, orally, once daily for up to 10 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, tablets, orally, once daily for 8 weeks, followed by vortioxetine placebo-matching tablets, orally, once daily for 2 weeks.
  Interventions: Drug: Vortioxetine; Drug: Placebo
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, tablets, orally, once daily for 8 weeks, followed by vortioxetine placebo-matching tablets, orally, once daily for 2 weeks.
  Interventions: Drug: Vortioxetine; Drug: Placebo
- Vortioxetine 20 mg (Experimental): Vortioxetine 10 mg, tablets, orally, once daily for 1 week, followed by vortioxetine 20 mg, tablets, orally, once daily for 7 weeks, followed by vortioxetine placebo-matching tablets, orally, once daily, for 2 weeks.
  Interventions: Drug: Vortioxetine; Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 10 mg; Vortioxetine 20 mg; Vortioxetine 5 mg
Drug: Placebo — Vortioxetine placebo-matching tablets

SUMMARY:
The purpose of this study is to assess the efficacy and safety of multiple doses of vortioxetine, once daily (QD), in participants with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took varying doses of vortioxetine.

The study enrolled 600 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 5 mg
* Vortioxetine 10 mg
* Vortioxetine 20 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in 14 countries in Europe and Asia. The overall time to participate in this study was up to 13 weeks. Participants made weekly visits to the clinic during the first 2 weeks of the 8-week treatment period and then every 2 weeks up to the end of the 8-week treatment period. Participants who completed the 8-week treatment period entered a 2-week discontinuation period to assess potential discontinuation symptoms 1 and 2 weeks after the end of the 8-week treatment period. A safety follow-up contact (visit or phone call) was made 4 weeks after completion of the 8-week double-blind treatment period (2 weeks after the end of the 2-week discontinuation period).

ELIGIBILITY:
Inclusion Criteria:

1. Suffers from Major Depressive Disorder as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.2x and 296.3x).
2. The reported duration of the current major depressive episode is at least 3 months at the Screening Visit.
3. Has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥26 at the Screening and Baseline Visits.
4. Has a Clinical Global Impression Scale-Severity (CGI-S) score ≥4 at the Screening and Baseline Visits.

Exclusion Criteria:

1. Has one or more of the following conditions:

   * Any current psychiatric disorder other than Major Depressive Disorder as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR; assessed by the Mini International Neuropsychiatric Interview: MINI). A participant who exhibits symptoms of anxiety is eligible unless fulfilling the diagnostic criteria for a current anxiety disorder per DSM-IV-TR.
   * Current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   * Current diagnosis or history of any substance-related disorder (except nicotine and caffeine-related disorders) as defined in the DSM-IV-TR. Participant with confirmed positive urine drug screens (except prescribed medications or a medication that does not constitute drug abuse) will be excluded.
   * Presence or history of a clinically significant neurological disorder (including epilepsy).
   * Neurodegenerative disorder. (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, etc.)
   * Any DSM-IV-TR axis II disorder that might compromise the study.
2. The current depressive symptoms of the participant are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
3. Has received electroconvulsive, vagal nerve stimulation, or repetitive transcranial magnetic stimulation therapy within 6 months prior to the Screening Visit.
4. Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
5. Is at significant risk of suicide or has a score ≥5 on Item 10 (suicidal thoughts) of the MADRS, or has attempted suicide within 6 months prior to the Screening Visit.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (70):
- Croatia (2):
  - Split, Croatia
  - Zagreb, Croatia
- Finland (4):
  - Helsinki, Finland
  - Kuopio, Finland
  - Oulu, Finland
  - Tampere, Finland
- Germany (10):
  - Berlin, Germany
  - Bochum, Germany
  - Chemnitz, Germany
  - Hanover, Germany
  - Leipzig, Germany
  - München, Germany
  - Nuremberg, Germany
  - Schwerin, Germany
  - Westerstede, Germany
  - Wiesbaden, Germany
- Hong Kong, Hong Kong, Hong Kong
- India (5):
  - Hyderabad, Andhra Pradesh
  - Ahmedabad, Gujarat
  - Kanpur, Uttar Pradesh
  - Lucknow, Uttar Pradesh
  - Varanasi, Uttar Pradesh
- Japan (9):
  - Tokoname-shi, Aichi-ken
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Omuta-shi, Fukuoka
  - Shirakawa-shi, Fukushima
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Tokyo, Tokyo
- Latvia (3):
  - Liepāja, Latvia
  - Riga, Latvia
  - Sigulda, Latvia
- Malaysia (2):
  - Johor Bahru, Malaysia
  - Kuala Lumpur, Malaysia
- Philippines (4):
  - Makati City, NCR
  - Mandaluyong, NCR
  - Manila, NCR
  - Quezon City, NCR
- Poland (5):
  - Bialystok, Poland
  - Gorlice, Poland
  - Leszno, Poland
  - Torun, Poland
  - Żuromin, Poland
- Romania (3):
  - Iași, Lasi
  - Târgu Mureş, Mureș County
  - Bucharest, Romania
- Russia (6):
  - Nizhny Novgorod, Russia
  - Rostov-on-Don, Russia
  - Saint Petersburg, Russia
  - Smolensk, Russia
  - Stavropol, Russia
  - Yekaterinburg, Russia
- Serbia (3):
  - Belgrade, Serbia
  - Kragujevac, Serbia
  - Senta, Serbia
- South Korea (4):
  - Sungnam-si, Gyeonggi-do
  - Incheon, Korea
  - Seoul, Korea
  - Yangsan, Korea
- Taiwan (4):
  - Changhua, Taiwan
  - Kaohsiung City, Taiwan
  - Taipei, Taiwan
  - Taoyuan Hsien, Taiwan
- Ukraine (5):
  - Chernigiv Region, Ukraine
  - Dnipropetrovsk, Ukraine
  - Kharkiv, Ukraine
  - Kiev, Ukraine
  - Luhansk, Ukraine

REFERENCES:
- [Derived] Adair M, Christensen MC, Florea I, Loft H, Fagiolini A. Vortioxetine in patients with major depressive disorder and high levels of anxiety symptoms: An updated analysis of efficacy and tolerability. J Affect Disord. 2023 May 1;328:345-354. doi: 10.1016/j.jad.2023.01.074. Epub 2023 Jan 26. PMID 36708956
- [Derived] Nishimura A, Aritomi Y, Sasai K, Kitagawa T, Mahableshwarkar AR. Randomized, double-blind, placebo-controlled 8-week trial of the efficacy, safety, and tolerability of 5, 10, and 20 mg/day vortioxetine in adults with major depressive disorder. Psychiatry Clin Neurosci. 2018 Feb;72(2):64-72. doi: 10.1111/pcn.12565. Epub 2017 Oct 3. PMID 28858412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 90 investigative sites in Japan, Europe and Asia/Oceania from 18 November 2010 to 25 April 2012.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 4 treatment groups, once a day placebo, 5 mg, 10 mg, or 20 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Started | 152 | 144 | 150 | 154
Treated | 152 | 144 | 148 | 150
Completed | 136 | 127 | 132 | 132
Not Completed | 16 | 17 | 18 | 22
Not completed — Pretreatment Event or Adverse Event (AE) | 6 | 2 | 9 | 9
Not completed — Major Protocol Deviation | 1 | 1 | 0 | 4
Not completed — Lost to Follow-up | 1 | 2 | 4 | 2
Not completed — Withdrawal of Consent | 3 | 9 | 3 | 4
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 2 | 2 | 2
Not completed — Noncompliance with Study Drug | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg | Total
Number analyzed (Participants) | 152 | 144 | 150 | 154 | 600
Age Continuous [Mean (Standard Deviation); unit: years] | 43.6 (11.57) | 44.2 (11.89) | 45.7 (10.90) | 44.0 (11.79) | 44.4 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 98 | 93 | 93 | 375
  Male | 61 | 46 | 57 | 61 | 225
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (or White, including Hispanic) | 104 | 101 | 104 | 105 | 414
  Asian | 48 | 43 | 46 | 49 | 186
Region of Enrollment [Number; unit: participants]
  Croatia | 0 | 1 | 0 | 2 | 3
  Finland | 5 | 5 | 5 | 5 | 20
  Germany | 50 | 50 | 50 | 49 | 199
  India | 3 | 3 | 3 | 2 | 11
  Japan | 33 | 32 | 31 | 33 | 129
  Latvia | 3 | 2 | 2 | 3 | 10
  Malaysia | 2 | 0 | 0 | 2 | 4
  Philippines | 4 | 2 | 4 | 3 | 13
  Poland | 20 | 18 | 20 | 21 | 79
  Romania | 5 | 4 | 6 | 3 | 18
  Russia | 13 | 13 | 12 | 13 | 51
  Serbia | 2 | 2 | 3 | 2 | 9
  South Korea | 6 | 6 | 7 | 8 | 27
  Ukraine | 6 | 6 | 7 | 8 | 27
Height [Mean (Standard Deviation); unit: cm] | 167.1 (8.75) | 167.2 (9.64) | 167.5 (9.40) | 167.5 (9.61) | 167.3 (9.33)
Weight [Mean (Standard Deviation); unit: kg] — Number of participants for whom weight data were available were 152, 144, 147 and 149 in each treatment group respectively.
  kg | 69.70 (16.901) | 70.57 (18.214) | 73.37 (19.014) | 70.21 (18.189) | 70.95 (18.095)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Number of participants for whom BMI data were available were 152, 144, 147 and 149 in each treatment group respectively.
  kg/m^2 | 24.82 (5.129) | 25.06 (5.432) | 25.93 (5.462) | 24.82 (5.206) | 25.15 (5.313)
Smoking Classification [Number; unit: participants]
  Current smoker | 51 | 50 | 50 | 56 | 207
  Ex-smoker | 22 | 19 | 21 | 11 | 73
  Never smoked | 79 | 75 | 79 | 87 | 320
History of Alcohol Consumption [Number; unit: participants]
  Never | 58 | 62 | 54 | 56 | 230
  Once monthly or less often | 52 | 41 | 54 | 53 | 200
  Once a week | 17 | 22 | 22 | 22 | 83
  2 to 6 times per week | 14 | 9 | 10 | 13 | 46
  Daily | 11 | 10 | 10 | 10 | 41
Status of Major Depressive Episode (MDE) [Number; unit: participants] — An MDE is a period marked by depressed mood, loss of interest or pleasure, disturbed sleep or appetite, low energy, feelings of guilt or low self-worth, and poor concentration.
  participants
    Single episode | 51 | 55 | 49 | 49 | 204
    Recurrent episode | 101 | 89 | 101 | 105 | 396
Pharmacotherapy for Current Major Depressive Episode [Number; unit: participants]
  Yes | 73 | 60 | 69 | 75 | 277
  No | 79 | 84 | 81 | 79 | 323
Montgomery Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  Number of participants for whom MADRS data were available were 152, 144, 147 and 149 in each treatment arm respectively.
  scores on a scale | 31.6 (3.56) | 31.6 (3.67) | 31.8 (4.02) | 31.7 (3.73) | 31.7 (3.74)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. Number of participants for whom CGI-S data were available were 152, 144, 147 and 149 in each treatment arm respectively.
  scores on a scale | 4.7 (0.66) | 4.7 (0.65) | 4.7 (0.66) | 4.7 (0.65) | 4.70 (0.65)
Sheehan Disability Scale (SDS) - Total score [Mean (Standard Deviation); unit: scores on a scale] — The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. Number of participants for whom SDS data were available were 132, 116, 119 and 121 in each treatment arm respectively.
  scores on a scale | 18.2 (5.28) | 17.9 (6.27) | 18.5 (5.42) | 18.2 (5.70) | 18.2 (5.65)
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity). Number of participants for whom HAM-A data were available were 152, 144, 148 and 150 in each treatment arm respectively.
  scores on a scale | 18.6 (6.83) | 18.9 (6.55) | 18.8 (6.66) | 18.5 (6.12) | 18.7 (6.53)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. Least squares (LS) means were from an Analysis of Covariance (ANCOVA) model with treatment as a fixed factor and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: The full analysis set included all randomized participants who received at least 1 dose of study drug. One patient in the placebo arm was excluded from all datasets due to enrollment in another clinical study. Only participants with Baseline and at least 1 post-baseline value are included. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 150 | 142 | 147 | 149
scores on a scale | -13.99 (0.783) | -14.61 (0.805) | -15.68 (0.791) | -15.82 (0.786)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; All statistical tests were 2-sided with the estimated P-values at the 5% level of significance; Test type: Superiority or Other; p = 0.9070, ANCOVA — Adjustment for multiplicity for the comparisons was based on the Dunnett-Hsu procedure; Analysis of covariance (ANCOVA), with treatment as a fixed factors and baseline MADRS as a covariate; LS Mean Difference = -0.61, 95% CI 2-sided [-3.258 to 2.035], Standard Error of Mean 1.123
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.3006, ANCOVA; Analysis of covariance (ANCOVA), with treatment as a fixed factors and baseline MADRS as a covariate; LS Mean Difference = -1.69, 95% CI 2-sided [-4.310 to 0.938], Standard Error of Mean 1.114
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.2399, ANCOVA; Analysis of covariance (ANCOVA), with treatment as a fixed factors and baseline MADRS as a covariate; LS Mean Difference = -1.82, 95% CI 2-sided [-4.436 to 0.794], Standard Error of Mean 1.110

2. Secondary Outcome: Percentage of Participants With a MADRS Response at Week 8
Description: Response is defined as a participant with a ≥50% decrease in Montgomery Åsberg Depression Rating Scale (MADRS) total score from Baseline. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Baseline and Week 8
Population: Full analysis set, only participants with Baseline and at least 1 post-baseline value are included. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 150 | 142 | 147 | 149
percentage of participants | 39.3 | 49.3 | 54.4 | 51.0

3. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 8
Population: Full analysis set, only participants with Baseline and at least 1 post-baseline value are included. LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 150 | 142 | 147 | 149
percentage of participants | 26.7 | 24.6 | 29.3 | 30.9

4. Secondary Outcome: Mean Clinical Global Impression Scale - Improvement (CGI-I) Score at Week 8
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from an ANCOVA model with treatment as a fixed factor and the Baseline Clinical Global Impression-Severity of Illness (CGI-S) score as a covariate.
Time Frame: Week 8
Population: Full analysis set, only participants with Baseline and at least 1 post-baseline value are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 150 | 142 | 148 | 150
scores on a scale | 2.54 (0.087) | 2.37 (0.089) | 2.27 (0.088) | 2.36 (0.087)

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and family life or home responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from an ANCOVA model with treatment as a fixed factor and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: Full analysis set, only participants with Baseline and at least 1 post-baseline value are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 126 | 109 | 114 | 118
scores on a scale | -6.20 (0.602) | -6.38 (0.647) | -7.97 (0.633) | -7.26 (0.622)

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event is defined as any AE whose onset occurs or intensity increases after the first dose of double-blind study medication through 2 weeks after the last dose of double-blind study medication.
Description: The safety analysis set included all patients who received at least 1 dose of study drug. One patient in the placebo arm was excluded due to enrollment in another clinical study. Any event spontaneously reported by the patient or observed by the investigator was recorded, irrespective of relation to study drug.
Arm/Group | Placebo | Vortioxetine 5 mg | Vortioxetine 10 mg | Vortioxetine 20 mg
Serious Adverse Events (participants affected / at risk) | 1/151 | 2/144 | 2/148 | 3/150
Other Adverse Events (participants affected / at risk) | 97/151 | 96/144 | 93/148 | 106/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 5 mg (N=144) | Vortioxetine 10 mg (N=148) | Vortioxetine 20 mg (N=150)
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Vortioxetine 5 mg (N=144) | Vortioxetine 10 mg (N=148) | Vortioxetine 20 mg (N=150)
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 3 | 2 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 11 | 26 | 27 | 37
Diarrhoea (Gastrointestinal disorders) | 14 | 7 | 6 | 5
Constipation (Gastrointestinal disorders) | 3 | 6 | 5 | 8
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 6 | 9
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Fatigue (General disorders) | 2 | 6 | 4 | 5
Thirst (General disorders) | 1 | 0 | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 18 | 24 | 18 | 21
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Headache (Nervous system disorders) | 21 | 16 | 19 | 23
Dizziness (Nervous system disorders) | 5 | 7 | 8 | 10
Hypoaesthesia (Nervous system disorders) | 4 | 1 | 1 | 1
Sedation (Nervous system disorders) | 1 | 2 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 4 | 4 | 9
Suicidal ideation (Psychiatric disorders) | 4 | 2 | 2 | 2
Depression (Psychiatric disorders) | 3 | 1 | 2 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5 | 4 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3
Somnolence (Nervous system disorders) | 2 | 7 | 7 | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.